CLINICAL TRIAL: NCT07049978
Title: Long-term Effect of Dupilumab on Acetylsalicylic Acid (ASA) Intolerance and Its Mechanisms in Patients With Non-steroidal Anti-inflammatory Drug-exacerbated Respiratory Disease (N-ERD)
Brief Title: Long-term Effect of Dupilumab in N-ERD
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Sven Schneider, MD, Priv.-Doz. DDr., Medical University of Vienna
Other Study IDs: DUPI-NERD-02
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: NSAID-Induced Asthma; NSAIDs Hypersensitivity; Chronic Rhinosinusitis (CRS); Asthma Bronchiale; Nasal Polyposis
MeSH Terms: conditions — Asthma, Aspirin-Induced; Nasal Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- N-ERD patients with long-term Dupilumab treatment: Patients diagnosed with N-ERD undergoing Dupilumab treatment between 3 and 4 years
  Interventions: Other: Observational follow-up of standard Dupilumab treatment

INTERVENTIONS:
Other: Observational follow-up of standard Dupilumab treatment — Patients undergoing Dupilumab treatment for N-ERD will be observed after three to four years of treatment to assess long term changes in ASA tolerance, clinical parameters, inflammatory biomarkers, quality of life, and nasal microbiome during ongoing treatment with Dupilumab. All participants are receiving Dupilumab as part of standard clinical care.

SUMMARY:
This prospective observational study investigates the long-term effects of Dupilumab in patients with NSAID-exacerbated respiratory disease (N-ERD). The study assesses changes in ASA tolerance, clinical parameters, inflammatory biomarkers, quality of life, and nasal microbiome during ongoing treatment with Dupilumab. All participants are receiving Dupilumab as part of standard clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Participated previously in our preliminary study (EK 1044/2020) and continued Dupilumab treatment since then. Long-term use of Dupilumab since the preliminary study will be assessed based on patient self-report, as there is currently no clinical test or laboratory parameter available to objectively verify treatment duration.
* Signed and dated informed consent has been obtained
* Current therapy with Dupilumab

Exclusion Criteria:

* Pregnancy (as determined by urine ß-HCG test)
* Clinically significant abnormal laboratory values and active infection (Tbc, HIV, hepatitis A/B/C)
* History of malignancy or immunodeficiency
* Chronic obstructive lung disorders (COPD), other obstructive lung disorders (bronchiolitis)
* Need for systemic corticosteroid therapy 1 month prior to screening visit
* Eosinophilic pneumonia and Churg-Strauss Syndrome
* Previous anaphylaxis and contraindications against ASA as outlined in the official prescribing information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with NSAID-exacerbated respiratory disease (NERD), previously included in a Dupilumab follow-up study, now being evaluated after ≥3 years of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in ASA tolerance | Historical (pre-treatment and 6 months) vs. current data (after ≥3 years of treatment)
  Change in aspirin tolerance assessed via oral provocation test with standardized protocol

SECONDARY OUTCOMES:
Change in Sino-Nasal Outcome Test 22 (SNOT-22) score compared to early response | Historical (pre-treatment and 6 months) vs. current data (after ≥3 years of treatment)
  Sinonasal symptoms assessed with SNOT-22 questionnaire at long-term follow-up, higher score means higher limitation by disease.
Change in European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3L) score compared to early response | Historical baseline and 6-month vs. current score (≥3 years post-treatment)
  General quality of life at long-term follow-up, higher score means good QoL.
Change in Asthma Control Questionnaire (ACQ-5) score | Historical baseline and 6-month vs. current score (≥3 years post-treatment)
  Asthma control evaluated via ACQ-5, high score means high disease burden.
Change in peripheral eosinophil count | Historical baseline and 6-month vs. current score (≥3 years post-treatment)
  Long-term effect of Dupilumab on peripheral eosinophils
Nasal microbiome composition at long-term follow-up | Historical baseline and 6-month vs. current score (≥3 years post-treatment)
  Microbial composition from nasal swabs assessed via sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Sven Schneider Dr. med. univ., MD, Principal Investigator — Senior doctor and Department of Otorhinolaryngology at Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schneider S, Poglitsch K, Morgenstern C, Quint T, Gangl K, Sinz C, Bartosik T, Campion NJ, Liu DT, Landegger LD, Tu A, Stanek V, Rocha-Hasler M, Bangert C, Eckl-Dorna J. Dupilumab increases aspirin tolerance in NSAID-exacerbated respiratory disease. Eur Respir J. 2023 Mar 16;61(3):2201335. doi: 10.1183/13993003.01335-2022. Print 2023 Mar. PMID 36549708